CLINICAL TRIAL: NCT07234123
Title: Conditioned Pain Modulation With Ultra-Brief Conditioning Stimulus
Brief Title: Cognitive Conditioned Pain Modulation
Acronym: CognitiveCPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Mayday Fund (Other)
Responsible Party: Principal Investigator, Hunter Hoffman, Research Scientist, University of Washington
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPM2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Conditioned Pain Modulation

STUDY DESIGN:
Intervention Model Description: within-subject design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single pain stimulus (Experimental): test pain stimulus alone
  Interventions: Behavioral: test stimulus
- dual pain stimuli (Experimental): simultaneous foot (test stimulus + wrist (conditioning stimulus)
  Interventions: Behavioral: conditioned pain modulation

INTERVENTIONS:
Behavioral: conditioned pain modulation — simultaneous stimuli to foot (test stimulus) and wrist (conditioning stimulus)
  Arms: dual pain stimuli
Behavioral: test stimulus — single brief stimulus to foot only
  Arms: Single pain stimulus

SUMMARY:
This "pain reduces pain" study looks at how the brain reduces pain when a person feels two painful sensations at the same time. There is considerable evidence that the brain can "turn down" pain using natural endogenous pain-control systems. The current CPM study measures whether attentional processes can also make a measurable contribution to pain inhibition alongside neurochemical mechanisms.

DETAILED DESCRIPTION:
Conditioned pain modulation (CPM) is a natural process where feeling pain in one part of the body (e.g., a conditioning stimulus to the wrist) can reduce pain felt in another part of the body (a test stimulus to the foot). There is considerable evidence from both animal and human studies that the painful conditioning stimulus can stimulate the brain to activate neurochemical pain-control pathways (e.g., endogenous opioids), which are believed to take 30-120 seconds to fully engage. The current CPM study measures whether attentional processes can also make a measurable contribution to pain inhibition alongside neurochemical mechanisms.

Primary measures: Graphic ratings scale "worst pain" ratings.

The primary measure of the current study graphic ratings scales (worst pain ratings) will measure how much pain participants feel on their foot during foot only (test stimulus), vs. how much pain participants feel on their foot (test stimulus during simultaneous foot (test stimulus) + wrist (conditioning stimulus).

The current investigators predict that pain (e.g., the conditioning stimulus) naturally demands attention and can pull attention away from the original pain source (the test stimulus), resulting in CPM-like reductions in pain of the test stimulus.

Secondary measure #1. Cognitive measures are introduced in the current study, to quantify how much (if at all) the conditioning stimulus reduces pain of the target stimulus via attentional mechanisms. Participants estimate what percentage of their attention was directed to their foot (the test stimulus) during foot only vs. during foot + wrist (test + conditioning stimulus). This will measure whether the conditiioning stimulus to the wrist reduces how much attention participants focus on their foot. Analyses will also measure whether the amount of attention shift away from the foot (via participants; subjective ratings) is correlated with CPM robustness (reduction in pain of foot during duel stimulation).

Secondary measure #2. As another secondary measure of attention during one vs. two simultaneous pain stimuli, this study involves a divided attention auditory listening task that becomes harder when pain demands more attention (Craik et al., odd number divided attention task during single test pain stimuli vs. simultaneous test + conditioning stimuli). The more errors the participant makes on the divided attention task, the more attention diverted away from the auditory task by pain. Analyses will measure whether the number of errors on the divided attention task is correlated with CPM robustness (reduction in pain of foot, during duel thermal stimulation).

Exploratory measures. As exploratory measures, participants will rate how distracted they were and how difficult it was to concentrate (on 0-10 rating scales during test stimulus alone verses test + conditioning noxious thermal heat stimuli).

In summary, embedding these cognitive measures into the CPM protocol may enhance mechanistic interpretation accuracy by quantifying attentional contributions to pain inhibition in specific CPM protocols, thereby complementing existing approaches to pain phenotyping and reducing unexplained variance in CPM outcomes.

ELIGIBILITY:
Inclusion criteria:

* Only University of Washington students in eligible psychological courses are
* eligible. General public is not eligible.
* Enrolled psychology students fluent in English,
* Age ≥18 y, able to follow instructions.

Exclusion criteria:

* Seizure history,
* Migraines,
* Diabetes,
* Extreme pain insensitivity,
* Motion sickness,
* or prior participation in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
worst pain ratings of foot only | rated immediately after each thermal stimulus
  graphic rating scale from 0 (no pain) to 10 (excruciating pain)
worst pain on graphic rating scale during test+conditioning stimulus | measured immediately after the stimuli
  graphic rating scale from 0 (no pain) to 10 (excruciating pain)

SECONDARY OUTCOMES:
% of attention devoted to foot during test stimulus only (0-100% scale) | rated immediately after the stimuli
  verbal ratings where higher numbers = more attention
% of attention devoted to foot during test+conditioning stimuli (0-100% scale) | rated immediately after the thermal stimuli
  verbal ratings where higher numbers = more attention
Divided attention during test stimulus only (% correct, where 100% is highest accuracy) | Day 1, during the thermal stimulus
  Accuracy monitoring a string of auditory numbers, the odd number task during test stimulus
Divided attention during test stimulus + conditioning stimulus (% correct, 100% is highest ) | Day 1, during the thermal stimuli
  Accuracy monitoring a string of auditory numbers, the odd number task during dual stimuli

OTHER OUTCOMES:
distraction difficulty during test stimulus only (0 to 10 scale, where 10 is most distracting) | immediately after the phase 1 thermal stimuli
  Exploratory: Distraction during the single test stimulus (graphic rating scales)
distraction difficult during simultaneous test + conditioning stimuli (graphic rating scale) | Exploratory: immediately after the phase 1 thermal stimuli
  Exploratory: 0-10 distraction during simultaneous test + conditioning stimulus (10 =highest distraction)
difficulty concentrating during test stimulus only (0 to 10 scale, 10 = most difficult concentr | Exploratory: immediately after the phase 1 thermal stimuli
  Exploratory: difficulty concentrating during the single test stimulus (graphic scales)
difficulty concentrating during simultaneous test + conditioning stimuli (graphic rating scale) | Exploratory: immediately after the phase 1 thermal stimuli
  Exploratory: difficulty concentrating during simultaneous test + conditioning stimulus, 10 = most difficult

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Hoffman, Principal Investigator — University of Washington
Locations (1):
- University of Washington Seattle, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Summary statistics will be made available to researchers upon reasonable request (e.g, for meta-analyses, etc). No individually identifiable information will be made available.
Time Frame: The de-identified summary data will be available from time of publication for at least five years after publication.
Access Criteria: The de-identified summary data will be e-mailed to researchers upon reasonable request

REFERENCES:
- [Background] Yarnitsky D. Conditioned pain modulation (the diffuse noxious inhibitory control-like effect): its relevance for acute and chronic pain states. Curr Opin Anaesthesiol. 2010 Oct;23(5):611-5. doi: 10.1097/ACO.0b013e32833c348b. PMID 20543676